CLINICAL TRIAL: NCT02290314
Title: Minimal Access Midline Lumbar Fusion Versus Traditional Open Posterior Lumbar Interbody Fusion for Degenerative Lumbar Spondylolisthesis
Brief Title: Midline Lumbar Fusion Versus Posterior Lumbar Interbody Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The London Spine Centre (Other)
Responsible Party: Principal Investigator, Dr. Christopher Bailey, Dr. Christopher Bailey, The London Spine Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105951
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Degenerative Lumbar Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- minimally invasive MID-line Lumbar Fusion (MIDLF) (Other): MIDLF surgery involves a minimally invasive midline laminectomy posterior approach to the lumbar spine. An incision that is smaller than the standard incision is made in the midline of the low back directly over the spinal levels. Afterward the pressure on the compressed nerves is released, and the disc between the affected vertebrae is completely removed. A metal cage filled with bone graft is placed as described in the PLIF procedure.
  Interventions: Procedure: minimally invasive MID-line Lumbar Fusion (MIDLF)
- posterior lumbar interbody fusion (PLIF) (Other): PLIF surgery involves a standard incision in the midline of the low back directly over the involved spinal levels. Afterward the pressure on the compressed nerves is released, and the disc between the affected vertebrae is completely removed. A metal cage filled with bone graft is placed in between the vertebral bodies where the disc usually lies. This will allow bone fusion (healing) to occur from one vertebral body to the other.
  Interventions: Procedure: Posterior lumbar interbody fusion (PLIF)

INTERVENTIONS:
Procedure: minimally invasive MID-line Lumbar Fusion (MIDLF)
  Arms: minimally invasive MID-line Lumbar Fusion (MIDLF)
Procedure: Posterior lumbar interbody fusion (PLIF)
  Arms: posterior lumbar interbody fusion (PLIF)

SUMMARY:
Degenerative lumbar spondylolisthesis is the forward displacement (slip) of one vertebra on an adjacent vertebra resulting in narrowing of the spinal canal or compression of the exiting nerve roots. It is commonly associated with low back and leg pain, and is a frequent reason for spine surgery particularly in individuals over age 65 years. Recently novel minimally invasive surgical techniques have heightened public and government interest by touting benefits of reduced approached-related morbidity which in turn leads to quicker recovery, shorter hospital stay, improved short-term clinical outcomes, and reduced health care cost. However, there is no randomized controlled trial evidence to describe the actual advantages and disadvantages associated with minimally invasive spinal fusion. This pilot study is a randomized control trial comparing minimally invasive MID-line Lumbar Fusion (MIDLF) to traditional "open" posterior lumbar interbody fusion (PLIF) with respect to length of stay, approach related morbidity, patient centered outcome measures, and cost-effectiveness in the treatment of degenerative lumbar spondylolisthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending Victoria Hospital
* Degenerative spondylolisthesis in the lumbar spine at one level
* Medically Suitable for surgical management
* Able to consent for surgery

Exclusion Criteria:

* Lytic spondylolisthesis
* Non degenerative stenosis: tumor, trauma
* Active infection
* On long term disability or workers compensation claims
* Drug or alcohol misuse
* Lack of permanent home residence
* Previous surgery in the lumbar spine at the surgical level
* Previous fusion in the lumbar spine
* Contraindication to surgery: medical co morbidities
* Unable to complete questionnaire: eg dementia
* Unable to give voluntary consent
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to discharge | Length of inhospital stay after surgery - average 4 days

SECONDARY OUTCOMES:
Approach-related in-hospital morbidity | At time of index surgery
  Blood loss, length of surgery, narcotic usage, nursing care, and adverse events will be compared between groups
Oswestry Disability Index | Enrollment, 6 weeks, 3 months, 6 months, 1 year, 2 year and 5 years
  The Oswestry Disability Index is an effective method of measuring disability in patients with back and leg pain and is well suited to patients who have had persistent severe disability. It is commonly utilized, validated and highly reproducible.
Cost-effectiveness of the two surgical approaches | Enrollment, 6 weeks, 3 months, 6 months, 1 year, 2 year and 5 years
  Economic score and cost analysis for each procedure

OTHER OUTCOMES:
Numeric rating scale for back pain intensity (0-10; 0=no pain; 10= worst pain) | Enrollment, 6 weeks, 3 months, 6 months, 1 year, 2 year and 5 years
Numeric rating scale for leg pain intensity (0-10; o=no pain; 10=worst pain) | Enrollment, 6 weeks, 3 months, 6 months, 1 year, 2 year and 5 years
General Health outcome measure (SF12) | Enrollment, 6 weeks, 3 months, 6 months, 1 year, 2 year and 5 years
  The SF12 is a standardized health related quality of life outcome questionnaire, which assesses 8 health domains. The physical and mental component can be derived. It has been validated and reliable when applied to the spine patient population
Patient satisfaction | Enrollment, 6 weeks, 3 months, 6 months, 1 year, 2 year and 5 years
  All things considered, how satisfied are you with the results of your recent treatment for your spine condition 1-7. This sentence is the recommended tool for assessing global satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bailey, Principal Investigator — London Health Sciences Centre and Western University
Locations (2):
- Canada (2):
  - London Health Science Centre, London, Ontario
  - London Health Sciences Centre, London, Ontario